CLINICAL TRIAL: NCT06161883
Title: Effect of the Intake of a Tomato Sofrito Preparation on Biomarkers of Cardiovascular Disease in an Overweight and/or Obese Population
Brief Title: Effect of Tomato Soffritto Intake on Biomarkers of Cardiovascular Disease in an Overweight and Obesity
Acronym: FRITOCARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ICCC-10 FRITOCARD; CEN-20101016 (Other Grant/Funding Number: CDTI-Spanish Ministry of Competitivity and Economy (MINECO))
Record Dates: First submitted 2023-11-20; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Dietary Exposure
Keywords: Dietary antiplatelet; Lipid profile; Endothelial activation; Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The intervention trial consisted of a single-center, prospective, controlled, randomized two-arm longitudinal crossover trial with a total duration of 16 weeks, which includes 2-weeks run-in period, 6 week intervention period (soffito or control group), 2-weeks wash-out period and 6 week intervention period (soffito or control group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soffritto group (Experimental): After a two-week run-in phase, participants (N=20) were randomly assigned to the Soffritto group. For 6 weeks, volunteers received soffritto (100 g/day). After the initial six-week phase, there was a two-week washout period, followed by a second six-week period in which participants were placed in the control group.
  Interventions: Other: Soffritto
- Control group (Experimental): After a two-week run-in phase, the participants (N=20) were randomly assigned to the control group. For 6 weeks, the volunteers did not receive any product. After the initial six-week run-in phase, there was a two-week washout period, followed by a second six-week period in which participants were switched to the Soffritto group (100g/day).
  Interventions: Other: Soffritto

INTERVENTIONS:
Other: Soffritto — The intervention trial was a single-center, prospective, controlled, randomized two-arm longitudinal crossover trial lasting 16 weeks. This duration encompassed a 2-week run-in period, a 6-week intervention period (either in the soffito or control group), a 2-week wash-out period, and another 6-week intervention period (soffritto or control group).
  Other Names: Tomato based products

SUMMARY:
The study is a prospective, controlled, randomized two-arm longitudinal crossover trial, performed in a single-centre. Hence, the investigators designed a clinical study aimed to investigate the effects of a daily intake of soffritto in overweight or obese class-1 individuals without other cardiovascular risk. After a run-in period of two-week, participants were randomly separated in two different intervention sequences (two-arms) of six-weeks in which volunteers were administered with a soffritto (100 g/day) or a control group (without soffritto). After the first six-week period, participants had a wash-out phase of two-week followed by a second six-week period in which groups exchanged their interventions. During the duration of the study, the volunteers were asked to maintain their usual diet, excluding raw or cooked tomatoes, as well as tomato-based products (sauces, ketchup, juices, etc.) other than those administered during the study in the corresponding periods.

DETAILED DESCRIPTION:
Sample size (N= 40) was calculated according results of previous studies on pigs (http://dx.doi.org/10.1016/j.trsl.2014.11.004). The study refers to healthy adult men (n=27) and women (n=13) with ages ranging from 25 to 60 years, non-smokers and with overweight (BMI: 25.0-29.9 kg/m2) or obesity class 1 (BMI: 30-34.9 kg/m2).

This study received approval from the Human Ethical Review Committee of Hospital Santa Creu I Sant Pau (Barcelona), with the reference number 12/181 and the date of approval being January 11, 2013. To confirm health status, all subjects underwent a complete physical examination conducted by the study physician.

The study lasted 16 weeks that were structured in:

* 2 weeks of run-in.
* 6 weeks of intervention period. During the intervention period, volunteers were administered with soffritto (100 g/day) or a control group (without soffritto).
* 2 weeks of wash-out.
* 6 weeks of intervention period. During the intervention period, volunteers exchanged their interventions

The volunteers visited the center at days 0, 14, 56, 70 and at the end of the intervention period (day 112).

Dietary habits were collected. Compliance was monitored by weekly telephone contact with participants and interviewing them at the end of each intervention period. Blood samples were collected early at the morning after twelve-hour fasting at baseline and at the end of each intervention phase. Blood samples were used for determining all variables of the study. Stool samples were obtained at baseline and after 42 days intervention for the study of platelet aggregation, lipid profile, biochemical measurements, vascular endothelial function and hemogram profile.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women 25-60 years of age
* BMI: >28 Kg/m2

Exclusion Criteria:

* Ischemic heart disease (and/or previous angina or AMI)
* Less than 25 years old and more than 60 years old
* Current/previous history of arrhythmia
* Cardiovascular co-morbidity (previous cardiovascular accidents and/or peripheral vascular disease)
* On current treatment with vasoactive drugs, fibrates or statins (see exception)
* Alcohol consumption of more than 60 gr/day
* Renal insufficiency (creatinine > 2 mg/dl)
* Presence of neoplasia
* Presence of systemic disease
* Psychiatric disease in treatment with psychotropic drugs
* Secondary dyslipidemia (nephrotic syndrome, hypothyroidism, others...)
* Being in a weight loss phase or expressing a desire for weight loss during the 3 months of the study duration.
* Having taken aspirin in the 10-day period prior to blood sampling.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03-15 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2014-02-28 (Actual)

PRIMARY OUTCOMES:
Changes from baseline of platelet aggregation (induced by different agonists: arachidonic acid [1 mM], collagen [2 and 5 µM] and ADP [5 and 20 µM] at day 42 | At days 0 and 42
  By the light transmission technique LTA. For all agonist results were expressed as the percentage of variation respect to the baseline value (100%).

SECONDARY OUTCOMES:
Changes from baseline of glucose levels at day 42 | At days 0 and 42
  Using routine commercially available assays
Changes from baseline of standard serum lipid profile (total cholesterol, high density lipoprotein-cholesterol, low density lipoprotein-cholesterol and triacylglycerols expressed as mg/dL) at day 42 | At days 0 and 42
  Routine commercially available assays were used for triglycerides, total cholesterol and high density lipoprotein cholesterol. Low density lipoprotein cholesterol was calculated using the Friedewald equation
Changes from baseline of vascular endothelial function (RHI, lnRHI, FRHI and AI@75) at day 42 | At days 0 and 42
  Digital plethysmography using the EndoPAT2000-device. Endothelial function was given as the reactive hyperaemia index (RHI) and the arterial stiffness as the augmentation index (AI) and AI standardized to a pulse of 75/min (AI@75). The natural logarithmically transformed RHI (lnRHI) values was also calculated. The Framingham RHI (FRHI) was calculated as the natural log-transformation of the RHI
Changes from baseline of hemogram profile at day 42 | At days 0 and 42
  Digital plethysmography using the EndoPAT2000-device
Changes from baseline of hemodynamic profile at day 42 | At days 0 and 42
  Blood pressure monitor (Sphygmomanometer)
Changes from baseline of hepatic enzymes (ALT, AST and GGT) at day 42 | At days 0 and 42
  Using routine commercially available assays
Changes from baseline of renal markers (creatinine, urea and uric acid) at day 42 | At days 0 and 42
  Using routine commercially available assays
Changes from baseline of BMI at day 42 | At days 0 and 42
  Dividing the body weight in kilograms by the square of height in meters (kg/m2)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Recerca-Hospital Santa Creu I Sant Pau, Barcelona, Spain